CLINICAL TRIAL: NCT02634424
Title: Interest of Preventive Personalized Treatment in Hemophilia A
Brief Title: PK Driven Prophylaxis for Hemophilia A
Acronym: OBTC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion and prophylaxy plateform being free to use for everyone in septembre 2016
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P140701
Record Dates: First submitted 2015-12-08; First posted 2015-12-18 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2016-08

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Prophylaxy; Pharmacokinetic; Bayesian
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MyPKFiT (Experimental): Personalized prophylaxis : Treatment is adjustment according to PK modeling
  Interventions: Device: MyPKFiT

INTERVENTIONS:
Device: MyPKFiT — Adjustment of the treatment dose using a decision support software according to the PK values
  Other Names: Personalized prophylaxis by PK modeling

SUMMARY:
The purpose of this study is to evaluate the implementation of pharmacokinetic (PK) driven prophylaxis in current clinical practice

DETAILED DESCRIPTION:
Starting from 3 pharmacokinetic (PK) points, data are entered in the PK calculator device, and treatment dose is adjusted following the results of PK values obtained and clinical bleeding data

ELIGIBILITY:
Inclusion Criteria:

* Male Patient
* Severe or moderately severe haemophilia A (FVIII = 2 %), preventively treated (processing) by ADVATE for at least 6 months,
* At last 6 years old,
* An informed consent must be signed by the patient or his legal representative for the patients minor.
* Affiliated to a national insurance scheme

Exclusion Criteria:

* Previous or actual treatment with FVIII inhibitors > 0,6 UB at the selection
* Induction of immune tolerance
* Planned orthopedic surgery for the 18 next months
* Any other haemostatic pathology
* Any treatment interacting on the haemostasis
* Patient under guardianship
* Patient participating in another biomedical research

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
Joint Annual Bleeding Rate | during 6 months before (retrospectively) and up to 12 months after using of myPKFiT
  Joint Annual Bleeding Rate assessed by usual patient book

SECONDARY OUTCOMES:
Total annual bleeding rate | during 6 months before (retrospectively) and up to 12 months after using of myPKFiT
  Total Annual Bleeding Rate assessed by usual patient book
Quality of life | up to 12 months
  Quality of life assessed by QoL-A-Haemo questionnaire for Adult and Haemo-QoL for children aged 6-17 years
Joint function | up to 12 months
  Joint function assessed thanks to score of joint state "Haemophilia Joint Health Score" (HJHS)
Adherence to treatment estimated as the quantity of Facteur VIII consumed reported to the prescribed quantity. | up to 6 and 12 months
  Quantity of Facteur VIII consumed will be assessed by usual patient book
Consumption of Factor VIII estimated by the Quantity of Facteur VIII consumed by thr patient. | during 6 months before (retrospectively) and up to 12 months after using of myPKFiT
  Consumption of Factor VIII assessed by usual patient book
Hemorrhagic Risk Sport | up to 6 and 12 months
  Hemorrhagic Risk Sport assessed by the scale "Hemophilia and sport"
Evolution between the annualized incidence of intercurrent events appeared or worsened under each treatment period (with and without myPKFit), globally, by System Organ ( SO) and Preferred Term ( PT) of the code MedDRA | during 6 months before (retrospectively) and up to 12 months after using of myPKFiT

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LAMBERT, MD, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France